CLINICAL TRIAL: NCT00813397
Title: Manageability and Safety Assessment of the SepraSpray Anti-adhesion Barrier in Abdominal Coelioscopic Surgery
Brief Title: Manageability and Safety Assessment of Sepraspray in Abdominal Surgery.
Acronym: C-MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSPRAY00608
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Adhesion Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sepraspray (Experimental): Receive Sepraspray
  Interventions: Device: Sepraspray
- Control (No Intervention): No Treatment, No Placebo

INTERVENTIONS:
Device: Sepraspray — Max. 10g of Sepraspray
  Arms: Sepraspray

SUMMARY:
This study will examine the performance of SeprasSpray in patients undergoing abdominal surgery (laparoscopic).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and over that require laparoscopic abdominal surgery

Exclusion Criteria:

* Patients who are pregnant or have an ongoing infectious complications from a previous surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (15):
- France (15):
  - CHU Amiens Nord, Amiens
  - Hopital Avicenne, Bobingy
  - Hopital Beaujon, Clichy
  - Centre Hospitalier Simone Veil, Eaubonne
  - Hopital Nord, Marseille
  - CHR Nantes-Hopital Hotel Dieu, Nantes
  - CHU Hopital de le'Archet, Nice
  - Institut Mutualiste Montsouris, Paris
  - CHU Bordeaux-Hopital du Haut Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Intercommunal de Poissy Saint-German, Poissy
  - CHU Charles Nicolle, Rouen
  - CHU Bordeaux Saint Andre, Talence
  - Hopital Purpan, Toulouse
  - CHU Hopital Trousseau, Tours

REFERENCES:
- [Derived] Berdah SV, Mariette C, Denet C, Panis Y, Laurent C, Cotte E, Huten N, Le Peillet Feuillet E, Duron JJ. A multicentre, randomised, controlled trial to assess the safety, ease of use, and reliability of hyaluronic acid/carboxymethylcellulose powder adhesion barrier versus no barrier in colorectal laparoscopic surgery. Trials. 2014 Oct 27;15:413. doi: 10.1186/1745-6215-15-413. PMID 25348087